CLINICAL TRIAL: NCT01325519
Title: A Prospective Randomized Trial Using Video Images in Advance Care Planning in Seriously Ill Hospitalized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010P002794
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Decision Making; Video Decision Aids
MeSH Terms: interventions — Decision Support Techniques; Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no intervention control group (No Intervention): control subjects
- experimental intervention group (Experimental): video decision aid viewed by subjects
  Interventions: Other: video decision aid

INTERVENTIONS:
Other: video decision aid — video
  Other Names: decision aid; film
  Arms: experimental intervention group

SUMMARY:
The purpose of this study is to compare the decision making of hospitalized subjects having a verbal discussion about CPR compared to subjects using a video.

DETAILED DESCRIPTION:
A.1. Aim 1: To recruit 150 subjects admitted to the inpatient general medicine ward with an overall prognosis of one year or less and randomly assign these subjects to: 1. a video visually depicting CPR preferences or 2. the current standard of care without the use of video (control).

Hypothesis 1: It is feasible to recruit and randomize 150 hospitalized subjects with an overall prognosis of one year or less.

A.2. Aim 2: To compare the care preferences for CPR and intubation among subjects randomized to video and subjects randomized to the current standard of care without the video.

Hypothesis 2: Subjects randomized to the video intervention will be significantly more likely to opt against CPR and intubation compared to those who do not see the video.

A.3. Aim 3: To compare code-status documentation in the electronic medical records between subjects randomized to the video and those who are receiving the current standard of care without the video.

Hypothesis 3: Subjects randomized to the video are more likely to have their code-status documented in the electronic medical records compared to those who do not see the video.

A.4. Aim 4: To compare the decisional conflict of subjects randomized to video and subjects randomized to the current standard of care without the video.

Hypothesis 4: When compared to subjects randomized to the current standard of care, subjects in the video intervention group will have lower decisional conflict (lower decisional conflict scores) when asked to choose CPR and intubation preferences.

A.5. Aim 5: To compare knowledge assessment of CPR of subjects randomized to video and subjects randomized to current standard of care without the video.

Hypothesis 5: When compared to subjects randomized to the current standard of care, subjects in the video intervention group will have higher knowledge assessment scores when asked questions regarding their understanding of CPR.

A.6. Aim 6: To compare code-status (CPR, and intubation) preferences in the electronic medical record on future hospitalizations up to one year post-hospital discharge of subjects randomized to video and subjects randomized to current standard of care without the video.

Hypothesis 6: Subjects randomized to the video are more likely to opt against CPR and intubation in the future compared to those who do not see the video.

ELIGIBILITY:
Inclusion Criteria

1. Over the age of 60
2. The ability to provide informed consent
3. The ability to communicate in English
4. And one of the following:

   1. An established diagnosis of metastatic cancer or
   2. An established diagnosis of advanced heart failure (NYHA class III/IV heart failure) or
   3. An established diagnosis of chronic obstructive lung disease with an FEV1 < 50% or
   4. Two hospitalizations within the last 6 months or
   5. An advanced illness or multiple comorbidities that are not otherwise specified with an overall prognosis of one year or less confirmed with the attending physician on service. Exclusion Criterion

1. Subject scores 6 or less on the Short Portable Mental Status Questionnaire, which is indicative of cognitive impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
preferences for medical care | within 48 hours of admission to the hospital
  preference for CPR

SECONDARY OUTCOMES:
knowledge of CPR | baseline and post-intervention
code status on subsequent admissions | subsequent hospital admissions

CONTACTS AND LOCATIONS:
Locations (1):
- MGH, Boston, Massachusetts, United States

REFERENCES:
- [Derived] El-Jawahri A, Mitchell SL, Paasche-Orlow MK, Temel JS, Jackson VA, Rutledge RR, Parikh M, Davis AD, Gillick MR, Barry MJ, Lopez L, Walker-Corkery ES, Chang Y, Finn K, Coley C, Volandes AE. A Randomized Controlled Trial of a CPR and Intubation Video Decision Support Tool for Hospitalized Patients. J Gen Intern Med. 2015 Aug;30(8):1071-80. doi: 10.1007/s11606-015-3200-2. Epub 2015 Feb 18. PMID 25691237